CLINICAL TRIAL: NCT06643663
Title: "Role of Guided Tissue Regeneration on Healing Outcome & Quality of Life in Combined Endo Perio Lesions With Communication: A Randomized Controlled Trial"
Brief Title: Role of GTR on Healing Outcome & Quality of Life in Combined Endo Perio Lesions With Communication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Parichay Singhal
Record Dates: First submitted 2024-05-22; First posted 2024-10-16 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Periapical Diseases; Endodontic Disease
Keywords: Guided tissue regeneration; healing; endo-perio lesions; endodontic surgery
MeSH Terms: conditions — Periapical Diseases; Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pt with apicomarginal defects & interproximal bone loss receiving GTR (Experimental): Surgery performed using ACM membrane and PRF plug.
  Interventions: Procedure: Endodontic Micro-Surgery
- Pt with apicomarginal defects & interproximal bone loss without GTR (Active Comparator): Surgery performed without ACM membrane and PRF plug.
  Interventions: Procedure: Endodontic Micro-Surgery

INTERVENTIONS:
Procedure: Endodontic Micro-Surgery — Surgery performed using ACM membrane and PRF plug in test group & without membrane & PRF in control group.

SUMMARY:
The recovery of periapical defects linked to periodontal communication frequently yields less satisfactory results. Numerous studies and case reports have highlighted the notable success achieved through the application of guided tissue regeneration techniques. More recently, autologous platelet concentrate plug & placental membrane have emerged as a treatment option for addressing such lesions. Nevertheless, there has been no study using PRF-Medium with ACM membrane on the healing of aforesaid lesion & quality of life assessment.

DETAILED DESCRIPTION:
RESEARCH QUESTION (PICO) Does the combined application of PRF-Medium plug and ACM membrane lead to superior healing outcomes compared to conventional technique in treating apico-marginal defects with interproximal involvement? AIM &OBJECTIVES: - AIM To assess whether the combined application of PRF-Medium and ACM membrane leads to improved healing outcomes and enhanced quality of life compared to conventional techniques in patients of apico-marinal defects with interproximal involvement. PRIMARY OBJECTIVE

1. To evaluate the impact of combined application of PRF-Medium and ACM membrane on healing outcomes in cases of apico-marginal defects with interproximal involvement with 2D periapical radiographs & 3D CBCT imaging. SECONDARY OBJECTIVE
2. To evaluate and compare differences in quality of life of patients after periapical surgery with use of PRF-Medium and ACM membrane in cases of apico-marginal defects with interproximal involvement. PICO P(Population)- Patients with non-vital teeth and persistant chronic suppurative apical periodontitis with apico-marginal defects and interproximal involvement. I(Intervention)-Endodontic surgery followed by placement of PRF-Medium plug and ACM membrane. C(Comparison)-Endodontic surgery without using any plug and membrane. O(Outcome)- Periapical healing after surgery in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age 16yrs and above.
2. Patients with apico-marginal defects and deep pocket upto apex of tooth.
3. Failed primary root canal treatment.
4. Presence of interproximal bone loss.
5. Negative response to vitality test.
6. ASA-1 or ASA- 2 according to the classification of the American Society of Anesthesiologists)

Exclusion criteria:

1. Presence of vertical root fracture
2. Presence of root perforations
3. ASA-3 or ASA-4 according to the classification of the American Society of Anesthesiologists)
4. Presence of root resorption
5. Combined endodontic-periodontic lesions.
6. Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Periapical healing assessment | Base line to 12 months
  Periapical healing comparison in 2 groups 2D radiographic healing by Rud et al and Molven et al criteria and 3D healing by modified PENN 3D Criteria. Healing will be categorised into complete, incomplete, uncertain, unsaisfactory.

SECONDARY OUTCOMES:
Quality of life assessment | Base line to 12 months
  to assess pain, swelling, mouth opening and effect on daily activities of patient among test and control group using OHIP-14 questionnaire. Pain Assesment with Value 0 indicate no pain & 100 indicate maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dr, Sanjay Tewari, MDS, Study Director — PGIDS, Rohtak, Haryana, 124001
Locations (1):
- Pgids Rohtak, Haryāna, India